CLINICAL TRIAL: NCT01389921
Title: Investigation of Lower Urinary Tract Afferent and Cortical Brain Activity During Lower Urinary Tract Stimulation Using Electroencephalogram Measurements
Brief Title: Study of Electroencephalogram (EEG) Measurement During Different Stimulations of the Lower Urinary Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulrich Mehnert (Other)
Collaborators: NCCR (National Center of Competence in Resaerch, Switzerland) (Network)
Responsible Party: Sponsor-Investigator, Ulrich Mehnert, Executive physician, University of Zurich
Organization: University of Zurich (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25/2009
Record Dates: First submitted 2011-06-28; First posted 2011-07-08 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Healthy; Nonneurogenic Neurogenic Bladder Dysfunction; Neurogenic Bladder Dysfunction Nos
Keywords: lower urinary tract; sensory evoked potential; contact heat evoked potential stimulation; electroencephalogram; cortical processing; bladder sensations; lower urinary tract dysfunction; overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy testpersons (Experimental): Electroencephalography recording during electrical stimulation of different locations of the lower urinary tract as well as during electrical and heat stimulation at the tibial and pudendal nerve and S3 dermatome.
  Interventions: Other: Electroencephalography
- patients with non-neurogenic OAB (Experimental): Electroencephalography recording during electrical stimulation of different locations of the lower urinary tract as well as during electrical and heat stimulation at the tibial and pudendal nerve and S3 dermatome.
  Interventions: Other: Electroencephalography
- patients with neurogenic OAB (Other): Electroencephalography recording during electrical stimulation of different locations of the lower urinary tract as well as during electrical and heat stimulation at the tibial and pudendal nerve and S3 dermatome
  Interventions: Other: Electroencephalography

INTERVENTIONS:
Other: Electroencephalography — Standard electroencephalography investigation according to the ICS standard Current recording of latency and amplitude of evoked potentials

SUMMARY:
The purpose of this study is to investigate afferent and cortical activities during bladder filling under different stimulations of the lower urinary tract. The participants of the study are healthy test persons and patients with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Written informed consent

Exclusion Criteria:

* Any psychological diseases
* Any renal, cardiac, and pulmonary diseases
* Pregnancy or breastfeeding
* Problems keeping calm for 60 minutes in the sitting position
* Medication influencing EEG or bladder function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Establishment of somatosensory evoked potentials of lower urinary tract stimulations | 3 times on an average period of three months
  EEG recording during electrical stimulation of different locations of the lower urinary tract as well as during electrical and heat stimulation at the tibial and pudendal nerve and S3 dermatome.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Mehnert, Dr., Principal Investigator — Neuro-Urology, Spinal Cord Injury Center & Research, University of Zürich, Balgrist University Hospital
Locations (1):
- Spinal Cord Injury & Research, University of Zürich, Balgrist University Hospital, Zurich, Switzerland

REFERENCES:
- [Background] Gregorini F, Knupfer SC, Liechti MD, Schubert M, Curt A, Kessler TM, Mehnert U. Sensory evoked potentials of the bladder and urethra in middle-aged women: the effect of age. BJU Int. 2015 Apr;115 Suppl 6:18-25. doi: 10.1111/bju.13066. PMID 25626360
- [Background] Knupfer SC, Liechti MD, Gregorini F, De Wachter S, Kessler TM, Mehnert U. Sensory function assessment of the human male lower urinary tract using current perception thresholds. Neurourol Urodyn. 2017 Feb;36(2):469-473. doi: 10.1002/nau.22956. Epub 2016 Jan 15. PMID 26773330
- [Background] Gregorini F, Wollner J, Schubert M, Curt A, Kessler TM, Mehnert U. Sensory evoked potentials of the human lower urinary tract. J Urol. 2013 Jun;189(6):2179-85. doi: 10.1016/j.juro.2012.11.151. Epub 2012 Nov 30. PMID 23206421